CLINICAL TRIAL: NCT02539537
Title: A Randomized Phase III Trial Comparing Chemotherapy With Folfirinox to Gemcitabine in Locally Advanced Pancreatic Carcinoma
Brief Title: A Randomized Phase III Trial Comparing Folfirinox to Gemcitabine in Locally Advanced Pancreatic Carcinoma
Acronym: NEOPAN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRODIGE 29 (UCGI 26); 2014-003510-82 (EudraCT Number)
Record Dates: First submitted 2015-08-03; First posted 2015-09-03 (Estimated); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Pancreatic Cancer; Carcinoma
Keywords: locally advanced pancreatic carcinoma; FOLFIRINOX
MeSH Terms: conditions — Pancreatic Neoplasms; Carcinoma | interventions — Gemcitabine; Leucovorin; Oxaliplatin; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Gemcitabine (Active Comparator): Gemcitabine 1000 mg/m² IV infusion over 30 minutes on D1 of each week for the 4 weeks of the first cycle (1 cycle = 4 weeks). For the following five cycles, gemcitabine infusion on D1, D8, and D15 of each cycle, followed by 1 week without injection (i.e. in total 4 cycles over 24 weeks; with 19 administrations of Gemcitabine).
  Interventions: Drug: Gemcitabine
- Arm B: Folfirinox (Experimental): Administered once every 14 days for 24 weeks (12 cycles). A cycle equals 14 days with injection on D1 of each cycle. Treatment starts with oxaliplatin (85 mg/m²) administration; IV infusion over 2 hours, followed by the simultaneous administration (using a Y-tubing) of folinic acid 400 mg/m² (racemic) (or 200 mg/m² if L-folinic acid) IV infusion over 2 hours and irinotecan 180 mg/m² IV infusion over 90 minutes. The irinotecan will begin 30 minutes after the start of the folinic acid infusion.
  5-Fluoro-uracil (5-FU) IV 2,400 mg/m²/h will be administered over 46 hours after the end of the folinic acid infusion, i.e. 1200 mg/m²/day for the duration of 2 days.
  Treatment will be continued for 24 weeks (12 cycles).
  Interventions: Drug: Folinic Acid; Drug: 5-Fluoro-uracil; Drug: Oxaliplatin; Drug: Irinotecan; Drug: L-folinic

INTERVENTIONS:
Drug: Gemcitabine
  Arms: Arm A: Gemcitabine
Drug: Folinic Acid
  Arms: Arm B: Folfirinox
Drug: 5-Fluoro-uracil
  Arms: Arm B: Folfirinox
Drug: Oxaliplatin
  Arms: Arm B: Folfirinox
Drug: Irinotecan
  Arms: Arm B: Folfirinox
Drug: L-folinic
  Arms: Arm B: Folfirinox

SUMMARY:
French national multicentric phase III trial evaluating chemotherapy with Folfirinox or gemcitabine in locally advanced pancreatic carcinoma.

DETAILED DESCRIPTION:
Comparative interventional prospective phase 3, randomized, open-label, multicentric trial comparing chemotherapy with Folfirinox to Gemcitabine in locally advanced pancreatic carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed adenocarcinoma of the pancreas
2. Proven unresectability after multidisciplinary discussion involving radiologist and a surgeon
3. Locally advanced (i.e.: no metastasis or suspicion of metastasis) and unresectable tumors: for example mesenteric or portal vein involvement, or > 180° encasement of the superior mesenteric artery, or celiac abutment (NCCN 2012 criteria)
4. Measurable tumor lesions with longest diameter ≥ 20 mm using conventional techniques or ≥ 10 mm with spiral CT scan according RECIST 1.1
5. WHO Performance status (PS) 0-1
6. Age ≥18 years
7. Patient with organ function as follows:

   * Absolute neutrophil count (ANC) ≥ 1.5 x 10⁹/L
   * Hemoglobin ≥ 10 g/dL
   * Platelets (PTL) ≥ 75 x 10⁹/L
   * Aspartate aminotransferase (AST) / alanine aminotransferase (ALT) ≤ 2.5 x upper limit of normal (ULN)
   * Bilirubin ≤ 1.5 x ULN
   * Creatinine ≤ 2 x ULN
   * Albumin > 0.75 x lower limit of normal (LLN)
   * Urea ≤ 2 x ULN
8. Adequate vital functions
9. Patient of child-bearing potential (for female patient: study entry after a menstrual period and a negative pregnancy test) must agree to use medically acceptable methods of contraception during the study and for 4 months after the last intake of study treatment for women and for 6 months after for men.
10. Patient information and signed informed consent form
11. Public or private health insurance coverage
12. Uracilemia < 16 ng/ml

Exclusion Criteria:

1. Patient treated for a cancer other than pancreatic cancer within 5 years before enrolment, with the exception of basal cell carcinoma or in situ cervical cancer
2. Patient with metastasis or with history of metastasis
3. Patient with grade III/IV cardiac problems as defined by the New York Heart Association Criteria. (i.e. congestive heart failure, myocardial infarction within 6 months before baseline)
4. Major comorbidity, active infection (HIV or chronic hepatitis B or C) or uncontrolled diabetes that may preclude the delivery of the treatment
5. Pre-existing neuropathy (Grade ≥ 2), Gilbert's disease or genotype UGT1A1 * 28 / * 28
6. Pregnant woman
7. Fructose intolerance
8. Patients currently treated by warfarin
9. Persons deprived of liberty or under guardianship
10. Psychological condition, family-, sociological- or geographical situation potentially hampering compliance with the study protocol and the follow-up schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2015-10-23 (Actual); Primary Completion 2022-02 (Actual); Study Completion 2023-09-25 (Actual)

PRIMARY OUTCOMES:
Progression-Free-Survival (PFS) | From randomization until disease progression or date of death, assessed up until to 128 weeks
  To compare Progression-Free-Survival (PFS) between the two treatment arms

SECONDARY OUTCOMES:
Composite index for treatment early severe toxicity | First four chemotherapy cycles, 16 weeks
  Biliary tract infection Grade 3-4 + any grade 5 toxicities + chemotherapy interruption for toxicity during the first four cycles.
Adverse events (NCI-CTCAE version 4.0); observance of chemotherapy | During treatment phase, 24 weeks
  Observance of chemotherapy
Overall Survival | Until death, assessed up 128 weeks after randomization
  The overall survival is the length of time from randomization that patients enrolled in the study are still alive. The outcome is to evaluate whether SRBT improves overall survival compared to standard of care.
Progression-free survival: pattern of failure | Until Disease Progression, assessed uo until 128 weeks after randomization
  The progression-free survival is the length of time during and after the treatment of a disease that a patient lives with the disease but it does not get worse.
Percentage of secondarily curative-intent surgery | Until surgery, if applicable, up until 128 weeks after randomization
  Percentage of patients who will undergo an exeresis of their pancreatic tumor, with R0 resection confirmed by anatomopathic pathology.
Objective tumour response, disease control and their duration | Until disease progression or date of death, assessed up until 128 weeks after randomization
  Objective tumour response, disease control and their duration (RECIST version 1.1),
Time to treatment failure | From randomisation to the end of treatment
  Time to treatment failure
Quality of life questionnaire - Core 30 (QLQ-C30) | assessed up until 128 weeks after randomization
  Developed by the EORTC, this self-reported questionnaire assesses the health-related quality of life of cancer patients in clinical trials. The questionnaire includes five functional scales (physical, everyday activity, cognitive, emotional, and social), three symptom scales (fatigue, pain, nausea and vomiting), a health/quality of life overall scale, and a number of additional elements assessing common symptoms (including dyspnea, loss of appetite, insomnia, constipation, and diarrhea), as well as, the perceived financial impact of the disease. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.

CONTACTS AND LOCATIONS:
Overall Officials: Michel DUCREUX, Professor, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (45):
- France (45):
  - Centre Hospitalier Intercommunal Aix-Pertuis, Aix-en-Provence
  - CHU Amiens - Hôpital Nord, Amiens
  - CHU d'Angers, Angers
  - Centre hospitalier d'Auxerre, Auxerre
  - Centre hospitalier Henri Duffaut, Avignon
  - Hôpital Avicenne, Bobigny
  - Institut Bergonié, Bordeaux
  - Polyclinique Bordeaux Nord, Bordeaux
  - CH Boulogne sur Mer, Boulogne-sur-Mer
  - CHU Côte de Nacre, Caen
  - Centre François Baclesse, Caen
  - Hôpital Trousseau, Chambray-lès-Tours
  - Hôpitaux civils de Colmar, Colmar
  - CH de Dijon, Dijon
  - CHD Vendée, La Roche-sur-Yon
  - Centre Hospitalier de Laon, Laon
  - Centre Oscar Lambret, Lille
  - CHU de Limoges, Limoges
  - Hôpital Edouard Herriot - Lyon, Lyon
  - Hôpital Saint Joseph Saint Luc, Lyon
  - Hôptal Européen, Marseille
  - Hôpital De La Timone, Marseille
  - Centre Hospitalier de Meaux, Meaux
  - Groupe Hospitalier du Havre Jacques Monod, Montivilliers
  - CHU Hotel Dieu, Nantes
  - Centre Antoine Lacassagne, Nice
  - CHR d'Orléans La Source, Orléans
  - Hôpital Saint Antoine, Paris
  - Groupe hospitalier Paris Saint Joseph, Paris
  - Groupe hospitalier Pitié Salpétrière, Paris
  - CH Annecy Genevois, Pringy
  - CHU - Robert Debre, Reims
  - CHU Rouen, Rouen
  - CHI Elbeuf, Saint-Aubin-lès-Elbeuf
  - Hôpital Privé des Côtes d'Armor, Saint-Brieuc
  - Centre Regional René Gauducheau, Saint-Herblain
  - Clinique mutualiste de l'Estuaire, Saint-Nazaire
  - Institut de cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez
  - Hôpital privé Saint Claude, Saint-Quentin
  - Centre Hospitalier de Soissons, Soissons
  - Centre Hospitalier de Saint Malo, St-Malo
  - Centre Paul Strass, Strasbourg
  - Polyclinique de l'Ormeau-GROP, Tarbes
  - Centre Hospitalier de Rangueil, Toulouse
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Yes
Unicancer will share de-identified individual data that underlie the results reported. A decision concerning the sharing of other study documents, including protocol and statistical analysis plan will be examined upon request.
Supporting Information: Study Protocol, SAP
Time Frame: The data shared will be limit to that required for independent mandated verification of the published results, the applicant will need authorization from Unicancer for personal access, and data will only be transferred after signing of a data access agreement.
Access Criteria: Unicancer will consider access to study data upon written detailed request sent to Unicancer, from 6 months until 5 years after publication of summary data.

REFERENCES:
- [Derived] Ducreux M, Desgrippes R, Rinaldi Y, Di Fiore F, Guimbaud R, Evesque L, Bachet JB, Vanelslander P, Lecomte T, Capitain O, Parzy A, Bolliet M, Etienne PL, Forestier J, El Hajbi F, Bignon AL, Lebrun-Ly V, De Sousa Carvalho N, Texier M, Bouche O. PRODIGE 29-UCGI 26 (NEOPAN): A Phase III Randomized Trial Comparing Chemotherapy With FOLFIRINOX or Gemcitabine in Locally Advanced Pancreatic Carcinoma. J Clin Oncol. 2025 Jul 10;43(20):2255-2264. doi: 10.1200/JCO-24-02210. Epub 2025 May 16. PMID 40378359